CLINICAL TRIAL: NCT01769573
Title: A First-in-Human Safety and Dose-Finding Study of New Type-16 Human Rhinovirus (RG-HRV16) Inoculum in Healthy Volunteers
Acronym: UWI-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2012-1036; IND15328 (Other: FDA)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: normal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 100 TCID50 (Experimental): RG-HRV16 dose of 100 TCID50 administered intranasally (0.25ml per nostril) one time.
  Interventions: Biological: RG-HRV16
- 1,000 TCID50 (Experimental): RG-HRV16 dose of 1,000 TCID50 administered intranasally (0.25ml per nostril) one time.
  Interventions: Biological: RG-HRV16
- 10,000 TCID50 (Experimental): RG-HRV16 dose of 10,000 TCID50 administered intranasally (0.25ml per nostril) one time.
  Interventions: Biological: RG-HRV16
- Placebo (Placebo Comparator): Diluent administered intranasally (0.25ml per nostril) one time.
  Interventions: Drug: Placebo
- 500 TCID50 (Experimental): RG-HRV16 dose of 500 TCID50 administered intranasally (0.25ml per nostril) one time.
  Interventions: Biological: RG-HRV16

INTERVENTIONS:
Biological: RG-HRV16 — A suspension of the RG-HRV16 virus in Minimal Essential Media (MEM, HyClone) containing 0.1% Human Serum Albumin
  Other Names: Rhinovirus type 16
  Arms: 1,000 TCID50; 10,000 TCID50; 100 TCID50; 500 TCID50
Drug: Placebo — The placebo to be used will be Minimal Essential Media (MEM, HyClone) containing 0.1% Human Serum Albumin. Placebo will be supplied in 2 ml borosilicate glass vials sealed with butyl stoppers containing 0.5 ml.
  Arms: Placebo

SUMMARY:
This research study will test different doses of RG-HRV16 to find the minimum dose needed to give research subjects cold symptoms of at least moderate intensity. The study will also test the safety of RG-HRV16. This information will be used in future studies (for example, to test antiviral preparations, sprays that could protect from getting a cold or decrease cold symptoms or to understand more about how rhinovirus can lead to asthma worsening). RG-HRV16 is a common cold virus that has been made in a new way and has not been used in humans before.

DETAILED DESCRIPTION:
Rhinoviruses are the most frequently cause of the common cold. HRV16 (Family Picornaviridae Genus Rhinovirus type 16) has been used extensively to induce colds in studies of experimentally inoculated volunteers that are designed to study the pathogenesis of colds and effects of antiviral medications.

Experimental inoculation with human rhinovirus type 16 (HRV16) administered intranasally via aerosolization has been used at the University of Wisconsin for over 30 years, and has proven to be a safe tool to reproducibly induce symptomatic colds. HRV has been linked with exacerbations of asthma and COPD, and this model has been used to evaluate inflammatory mechanisms and to test the efficacy of treatments for the common cold. Recent refinements in the technology available to produce and safety test reagents that are intended to be administered to human volunteers as part of research protocols has prompted us to produce a new lot of HRV16 in accordance with standards of current Good Manufacturing Procedures (cGMP). For this inoculum, we have used a cDNA clone (reverse genetics) to generate source virus, thus this new virus inoculum will be referred to as RG-HRV16.

This approach has two main advantages over using viruses isolated from nasal secretions. First, several "new" respiratory viruses (e.g. metapneumovirus, bocavirus, SARS, rhinovirus group C) have been discovered in the past 10 years, and there is little doubt that additional viruses will be discovered. Therefore, it is impossible to ensure that nasal secretions that are chosen for isolation of "seed virus" contain only the pathogen of interest. This problem is minimized through the use of virus derived from a cDNA clone that was produced in E. coli. Second, RNA viruses, such as HRV, mutate as the virus grows because their RNA polymerases have no error-correcting function. The cDNA clone, reproduced by the much more accurate E. coli DNA polymerase, provides a stable source of virus sequence for production of future inocula.

This study represents a first-in-human, phase 1 study to assess the safety of RG-HRV16 in humans and identify the dose needed to produce moderate-to-severe colds in 75% of HRV16-seronegative human volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to grant written informed consent (in English) and cooperate with study procedures and requirements including willingness to avoid cold symptom medications during the study.
2. Age between 18 and 50 years (children and older adults will be excluded from the study due to the possibility of greater morbidity associated with upper respiratory infections in these age groups).
3. Absence of HRV16 neutralizing antibody.
4. Safety laboratory assessments within normal University of WI Hospital and Clinics (UWHC) ranges or grade 1 (mild) laboratory abnormalities which are deemed not clinically significant in the judgment of the PI. Labs to include CBC with differential and platelets, BUN, creatinine, AST, ALT and IgA and IgG serum immunoglobulins. Any lymphopenia outside of the normal range will be an absolute exclusion.
5. Subjects must be willing to refrain from taking nasal decongestants, antihistamines or cough/cold preparations (this includes dietary supplements and homeopathic preparations used specifically for cold/flu e.g., vitamin C, zinc, echinacea) within the 7 days prior to Visit 1 and throughout the study until after the completion of Visit 5.

Exclusion Criteria:

1. A chronic medical condition, which may increase risk or interfere with the conduct of the study, including, but not limited to heart disease, Type I of II diabetes mellitus, asthma, COPD, other chronic lung disease, perennial rhinitis and chronic rhinosinusitis.
2. Subjects with household contacts who are pregnant or planning a pregnancy during the main subject's participation, who have chronic respiratory disease, who are children under the age of 2 years, or who are adults over 50 years of age.
3. Subjects who provide healthcare services or work with elderly or children (e.g. daycare provider, senior citizen care giver).
4. Subjects with seasonal allergies will be excluded only if allergy symptoms are present at baseline, or are anticipated to occur during the study period.
5. Smoking within the past 6 months.
6. Subjects who have received immunosuppressive treatment within the last 12 months.
7. Upper respiratory infection (URI or sinusitis) in the past 4 weeks.
8. Subjects with a history of a significant adverse reaction or intolerance to a previous live, attenuated vaccine.
9. Pregnant or breastfeeding women or a woman who has a planned pregnancy during the course of the study.
10. Unwillingness of study participants to use adequate birth control methods during the course of the study. Adequate birth control methods include oral contraceptives, injections such as Depo-Provera, an intrauterine device or double-barrier contraception (combination of condom and contraceptive sponge or cervical cap and spermicide or another combination approved in writing by the Principal Investigator).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Gern, MD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo
Started | 10 | 6 | 10 | 0 | 10
Completed | 10 | 6 | 10 | 0 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The trial completed and reached its goal without needing to enroll into the 10,000 TCID50 group.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo | Total
Number analyzed (Participants) | 10 | 6 | 10 | 0 | 10 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 10 | 0 | 10 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 6 | 0 | 9 | 26
  Male | 2 | 3 | 4 | 0 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 9 | 5 | 10 | 0 | 10 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 4 | 8 | 0 | 10 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 10 |  | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Colds With at Least Moderate Intensity
Description: The percentage of colds of at least moderate intensity examined by RG-HRV16 dose; this will be measured by the number of subjects per RG-HRV16 dose group who have maximum weekly cold symptom score of ≥7 out of 39 on the modified Jackson criteria during the first week after inoculation
Time Frame: 1 week
Population: The trial completed and met its goal before needing to enroll into the 10,000 TCID50 group.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo
Number analyzed (Participants) | 10 | 6 | 10 | 0 | 10
Participants | 4 | 2 | 7 | 0 | 0

2. Primary Outcome: Frequency of Adverse Events
Description: Safety as determined by the frequency of adverse event reporting examined by RG-HRV16 dose.
Time Frame: 4 weeks
Population: The trial completed and met its goal before needing to enroll into the 10,000 TCID50 group.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo
Number analyzed (Participants) | 10 | 6 | 10 | 0 | 10
Participants | 4 | 1 | 5 | 0 | 3

3. Secondary Outcome: Mean Cold Symptom Score
Description: The Mean Cold Symptom Score induced by each RG-HRV16 dose and by the placebo inoculation. The scale is called the Jackson Criteria for Cold Symptom Assessment. There are 13 variables of cold symptoms that each participant scores 0 (not present), 1 (mild), 2 (moderate) to 3 (severe), twice per day, once at 8am and once at 8pm. The 13 variables are: cough, nasal discharge, sneezing, stuffy nose, sore throat, headache, malaise, chilliness, shaking chills, fever, laryngitis, aching joints or muscles, and watery/burning eyes. The scores are added up for each time point, with a minimum score of 0 and a max score of 39 per time point. The highest score per day is taken and the highest score over the 7 day period starting from the day of the inoculation and for 7 days is deemed the mean cold symptom score. The higher the score, the more cold symptoms the participant reports and the worse the participant feels.
Time Frame: 4 weeks
Population: For the manuscript, the 500 TCID50 group was excluded from this analysis due to incomplete data that could not be analyzed appropriately.
  The trial completed and met its goal before needing to enroll into the 10,000 TCID50 group.
Measure: Mean (Standard Deviation); unit: peak symptom score
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo
Number analyzed (Participants) | 10 | 6 | 10 | 0 | 10
peak symptom score | 7.5 (5.0) | 7.3 (1.9) | 11.4 (7.8) |  | 1.9 (1.7)

4. Secondary Outcome: Infection Rate
Description: Infection rate per RG-HRV16 dose as measured by the percentage of individuals in the dosing group with detectable viral shedding.
Time Frame: 4 weeks
Population: The trial completed and met its goal before needing to enroll into the 10,000 TCID50 group.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo
Number analyzed (Participants) | 10 | 6 | 10 | 0 | 10
Participants | 10 | 6 | 10 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of signed consent until completion of study or roughly 60 days.
Description: No participants were enrolled in the 10,000 TCID50 group as the study met its goals early. All other groups report that all participants were at risk for Other Adverse Events, All-Cause Mortality and Serious Adverse Events.
Arm/Group | 100 TCID50 | 500 TCID50 | 1,000 TCID50 | 10,000 TCID50 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/10 | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/10 | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 1/6 | 5/10 | 0/0 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 TCID50 (N=10) | 500 TCID50 (N=6) | 1,000 TCID50 (N=10) | 10,000 TCID50 (N=0) | Placebo (N=10)
Headache (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Headache secondary to alcohol consumption
Migraine (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Migraine
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Headache after fall on ice
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Sinusitis
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Upper respiratory infection
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Muscle soreness secondary to skiing
IgA < 50 mg/dl (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — IgA < 50mg/dl
Heart rate < or equal to 54 (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Heart rate < or equal to 54
Heart rate > or equal to 101 (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) — Heart rate > or equal to 101
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dermatitis related to scented laundry detergent
Nasal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pain after nasal brush procedure
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Rash to bilateral inner elbow
Blepharitis to right eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Blepharitis to right eye, flare up
Crusted upper lip vesicle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Crusted upper lip ulceration (cold sore) ~ 1 cm diameter, a few intact vesicles
Lymph node swelling (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — R. anterior cervical lymph nodes swelling ~ 3 cm diameter

LIMITATIONS AND CAVEATS:
Limitations include inclusion of healthy adults as study subjects; it is possible that individuals with chronic respiratory disease (e.g. asthma, COPD) could develop milder colds and lower respiratory infections with lower doses of virus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes